CLINICAL TRIAL: NCT02258256
Title: Pilot Clinical Assessment of the Diagnostic Capability, Usability, and Function of an Automatic Blood Pressure Monitor for Use in the Diagnosis and Management of Pre-eclampsia in a Low-resource Hospital
Brief Title: Pilot Assessment of an Auto Blood Pressure Monitor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William Marsh Rice University (Other)
Collaborators: University of Malawi (Other)
Responsible Party: Principal Investigator, Rebecca Richards-Kortum, Stanley C. Moore Professor of Bioengineering, William Marsh Rice University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 14-082F-C; (COMREC) P.04/14/1548 (Other Grant/Funding Number: Merck for Mothers: 51262)
Record Dates: First submitted 2014-09-25; First posted 2014-10-07 (Estimated); Results first posted 2018-12-21 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Pre Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Intervention Model Description: Pregnant women will have their blood pressure measured by both the experimental device (Sphygmo ) and the gold-standard, commercial device (GE Dinamap Procare).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sphygmo (Experimental): All subjects will have blood pressure measured by both the research device (Sphygmo) and the commercially available device. All clinical decisions will be made using measurements from the commercially available device
  Interventions: Device: Sphygmo

INTERVENTIONS:
Device: Sphygmo — A team of engineers from Rice University has recently developed Sphygmo, an ambulatory, low-cost blood pressure monitor for use in the diagnosis and management of pre-eclampsia in low-resource hospitals

SUMMARY:
The purpose of the study is to help make a lower cost automatic blood pressure monitor device for diagnosis and monitoring of pre-eclampsia in pregnant women, where automatic blood pressure monitoring is limited or not available. The study will compare this low cost device to a commercially available system used for pre-eclamptic women in many United States hospitals that the investigators will be bringing to Malawi as a part of this study.

The team hopes to show that this lower cost blood pressure machine works well and can help women with pre-eclampsia. The study also aims to see if this machine is easy for the nurse to use.

20 women who are either at-risk or diagnosed with pre-eclampsia will be enrolled at Queen Elizabeth Central Hospital. First, a nurse will fit the test device cuff on one arm of the subject and the commercially available cuff on the opposite arm. A trained research assistant and the nurse will record the blood pressure measurements and document any alarm indications made by each device. Blood pressure measurements will continue until monitoring is no longer clinically prescribed.

The results of this study will help researchers understand the performance and usability of this device in Malawi and help decide if any design changes are needed.

DETAILED DESCRIPTION:
The research team at Rice University has developed Sphygmo, an automatic blood pressure monitor to be used for the monitoring and diagnosis of pre-eclampsia in pregnant women, particularly in low-resource settings where current blood pressure monitoring is limited. This study aims to evaluate the capabilities of the device in the setting for which it was designed - a low-resource hospital.

This study will compare the Sphygmo device to a commercially available automatic blood pressure monitor that is used in pre-eclamptic women. The main objective of this study is to determine whether the Sphygmo device correctly identifies instances where blood pressure measurement meets the diagnostic criteria for mild or severe pre-eclampsia during monitoring of at-risk mothers. Additionally, this study aims to understand the frequency and type of any complications associated with use of the Sphygmo in a resource-limited clinical setting.

The study will include 20 eligible and consenting women at QECH who are clinically identified as at-risk for pre-eclampsia or have already been diagnosed with pre-eclampsia by their doctors. All participants will undergo the same protocol (monitoring with both Sphygmo and the commercially available device). First, a nurse will fit a Sphygmo device cuff on one arm of the subject and the commercially available device cuff on the opposite arm. A trained research assistant will be continuously on hand to assist the nurse in the device setup and record the blood pressure measurements and any alarm indications made by each device. Blood pressure measurements by Sphygmo and the commercially available device will continue until monitoring is no longer clinically prescribed. In addition, blood pressure will be taken via clinical auscultatory measurement with a stethoscope and aneroid gauge at regular intervals. This third method will help us confirm the accuracy of the two devices. All clinical decisions will be made according to the commercially available device's measurements.

The key results of the study will be the ability of the Sphygmo device to identify blood pressure levels corresponding to mild and severe pre-eclampsia. Additionally, the investigators will document any user errors or device malfunction. These results will provide information on the performance and ease of use of the device and will also alert the research team of any necessary changes needed for the device.

ELIGIBILITY:
Inclusion Criteria:

* Women who have been identified as at-risk for pre-eclampsia or have been diagnosed with pre-eclampsia during a visit to QECH.
* Women who have been clinically identified to benefit from continuous blood pressure monitoring.
* Women ages 18 or older.

Exclusion Criteria:

* Pregnant women who have already developed eclampsia.
* Women under age 18.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca R Richards-Kortum, PhD, Principal Investigator — William Marsh Rice University; Ronald Mataya, MD, Principal Investigator — University of Malawi
Locations (1):
- Queen Elizabeth Central Hospital, Blantyre, Malawi

REFERENCES:
- [Background] Magee LA, Abalos E, von Dadelszen P, Sibai B, Easterling T, Walkinshaw S; CHIPS Study Group. How to manage hypertension in pregnancy effectively. Br J Clin Pharmacol. 2011 Sep;72(3):394-401. doi: 10.1111/j.1365-2125.2011.04002.x. PMID 21545480
- [Background] Wagner LK. Diagnosis and management of preeclampsia. Am Fam Physician. 2004 Dec 15;70(12):2317-24. PMID 15617295
- [Background] De Greeff A, Ghosh D, Anthony J, Shennan A. Accuracy assessment of the Dinamap ProCare 400 in pregnancy and preeclampsia. Hypertens Pregnancy. 2010 Jan;29(2):198-205. doi: 10.3109/10641950902968650. PMID 20367507
- [Background] Turner JA. Diagnosis and management of pre-eclampsia: an update. Int J Womens Health. 2010 Sep 30;2:327-37. doi: 10.2147/IJWH.S8550. PMID 21151680
- [Background] Dekker G, Sibai B. Primary, secondary, and tertiary prevention of pre-eclampsia. Lancet. 2001 Jan 20;357(9251):209-15. doi: 10.1016/S0140-6736(00)03599-6. PMID 11213110

RESULTS

PARTICIPANT FLOW:
Groups:
- Preeclamptic Women: All subjects are pre-eclamptic women who will have their blood pressure measured by both the research device (Sphygmo) and the commercially available device. All clinical decisions will be made using measurements from the commercially available device
  Sphygmo: A team of engineers from Rice University has recently developed Sphygmo, an ambulatory, low-cost blood pressure monitor for use in the diagnosis and management of pre-eclampsia in low-resource hospitals
Period: Overall Study
Arm/Group | Preeclamptic Women
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Preeclamptic Women
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 28 [20 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Malawi | 11

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Blood Pressure Measurement by Sphygmo Relative to the Clinical Standard.
Description: Mean systolic and diastolic pressures measured by the Sphygmo device blood pressure measurement and the commercially available device. Measurements were taken multiple times over the course of 24-72 hours at intervals determined by the supervising clinician. Mean blood pressure for each participant was measured using each device and compared between the two devices (Sphygmo minus Standard). The reported values represent the mean systolic and diastolic blood pressures measured by Sphygmo vs Gold Standard device, averaged across all participants
Time Frame: Measured during a single study visit, up to 24-72 hours.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Preeclamptic Women
Number analyzed (Participants) | 11
mmHg
  Systolic Mean BP - Sphygmo | 125.3 (31.8)
  Mean Diastolic BP - Sphygmo | 85.2 (29.8)
  Mean Systolic BP - GE Dinamap | 129.8 (24.8)
  Mean Diastolic BP - GE Dinamap | 76.9 (17.0)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the length of the subject visit (24-72 hours).
Arm/Group | Preeclamptic Women
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-06-25): https://cdn.clinicaltrials.gov/large-docs/56/NCT02258256/Prot_SAP_000.pdf